CLINICAL TRIAL: NCT06005090
Title: A Comparison of the Effects of Bicortical Locking and Far Cortical Locking Techniques on Clinical, Functional and Radiological Results During Minimally Invasive Plate Osteosynthesis of Tibial Distal Metaphyseal Fracture
Brief Title: Is Far Cortical Locking More Effective Than Bicortical Locking in Treating AO 43A1-3 Fractures?
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İsmail Demirkale, Clinical professor, Saglik Bilimleri Universitesi
Other Study IDs: 2012-KAEK-15/2103
Record Dates: First submitted 2023-08-04; First posted 2023-08-22 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Tibia Distal Fracture; Nonunion of Fracture of Tibia
Keywords: Extra-articular; distal tibia; MIPO; far cortical locking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FCL group: Plate fixation performed with the use of far cortical locking (2 point screw fixation into the plate and far cortex of the diaphysis)
  Interventions: Procedure: Far Cortical Locking Technique
- BL group: Traditional 3 point fixation of the screw into two cortices of the diaphysis and into the plate

INTERVENTIONS:
Procedure: Far Cortical Locking Technique — Apart from the traditional 3 point fixation of the locking screw this technique compromises two point fixation of the screw where one into the plate and the other is into the far cortex of the diaphysis. The near cortex was widened by 3.2 mm of dirll bit to eliminate the fixation of the screw into the near cortex
  Groups: FCL group

SUMMARY:
Delayed union or nonunion, which is a common complication of periarticular fractures repaired with angled locking plate systems, may be due to the unintentionally rigid formation of this system. This study aimed to compare the results of the treatment of distal tibial fractures made more flexible using the far cortical locking (FCL) technique with the classical bicortical locking screw (BL) technique.

DETAILED DESCRIPTION:
Extra-articular distal tibia fractures are uncommon; it constitutes less than 10% of all lower extremity fractures, but even if the fracture is closed, contusion and fracture blisters may accompany these fractures, which can be very effective in deciding the type of treatment because the soft tissue envelope surrounding the tibia is very thin. Discussions on the method of fixation of these fractures continue and seem to never end. Since comparative studies with two popular methods, intra-medullary nailing (IMN) and minimally invasive plate osteosynthesis (MIPO), eventually yielded similar results, the choice based on experience and patient-specific characteristics, described as surgeon comfort, has been more accepted.

Malunion after IMN is a common problem and may be caused by the gradual enlargement of the canal after the isthmus or the incomplete centering of the proximal insertion site of the nail. On the contrary, the most common complications reported after MIPO are delayed union, nonunion and infection. In the MIPO technique, angle-stable locked plates are used, which can prevent shear displacement and provide more than 0.2 mm of axial interfragmentary movement, allowing the formation of natural callus tissue. Different methods can be applied to make the partially rigid mechanical environment created by these plates more flexible. These can be diaphyseal fixation with conventional non-locking screws or far cortical locking (FCL), lengthening the bridging plate, or dynamizing the plate with active plates. The FCL method, which changes the axial load with the more parallel interfragmentary method and provides progressive symmetrical mineralization of the callus tissue, is based on the principle that a system that works like an external fixator but works as an internal fixator.

It is thought that this method, which can be defined biomechanically in this way, can prevent the formation of insufficient callus, which may occur especially between plate and bone, in the treatment of periarticular fractures. However, studies on this subject are insufficient in number. Therefore, we aimed to compare the radiological and clinical results of two different diaphyseal fixation models that we performed in the treatment of extra-articular distal tibial metaphyseal fractures with the MIPO method. Our hypothesis is that fixation with the FCL method will provide faster complete union compared to the classical locking plate technique, where the diaphyseal fixation is fixed at all three points with locking screws.

ELIGIBILITY:
Inclusion Criteria:

* closed extra articular AO 43A1-3 distal tibial fractures
* Skeletally mature patients
* giving informed consent
* competent neurological and vascular status

Exclusion Criteria:

* open fractures
* intraarticular extension,
* pathological fractures
* with poor medical health
* patients with deep abrasion or extensive skin contusion and crush injury preventing one-satge MIPPO

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature patients with closed extra articular AO 43A1-3 distal tibial fractures
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
RUST score | between 1.5, 6, 9th month and 12th month control
  Radiological Union Score of Tibia with a maximum of 12 points which means full union of all cortices

SECONDARY OUTCOMES:
AOFAS scores | between 1.5, 6, 9th month and 12th month control
  American Orthopedic Foot and Ankle Society scores range from 0 to 100, with healthy ankles receiving 100 points
Johner and Wruhs' Criteria | at 12th month control
  final functional evaluation of the ankle that includes the conditions of union and infection, as well as deformity and mobility, categorizes patients as excellent, good, fair, and poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Keçiören SUAM, Ankara, Turkey (Türkiye)